CLINICAL TRIAL: NCT05905692
Title: Evaluation of the Impact of L- Carnitine in Intradialytic Hypotension in Pediatric Patients on Regular Hemodialysis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Radwa Maher Abd El Kader El Borolossy, Lecturer of clinical pharmacy, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RHDIRB202011031 REC#154
Record Dates: First submitted 2023-05-29; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Intradialytic Hypotension
MeSH Terms: interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- L carnitine group (Experimental): patients will take L carnitine (20 mg/kg/day) 3 times per week (on the same days of the dialysis session, 30 minutes before the session)
  Interventions: Drug: L Carnitine
- Placebo group (Placebo Comparator): patients will take placebo 3 times per week (on the same days of the dialysis session, 30 minutes before the session)
  Interventions: Drug: L Carnitine

INTERVENTIONS:
Drug: L Carnitine — L carnitine will be given to group 1 (20 mg/kg/day) 3 times per week

SUMMARY:
Intradialytic hypotension (IDH) is defined as less than the 5th percentile of SBP measurements and is associated with clinical symptoms, such as abdominal pain, nausea, vomiting, muscle cramps, restlessness, light-headedness, syncope, and anxiety. In adults There is no consensus definition of IDH, however, according to the Kidney Disease Outcomes Quality Initiative and European Best Practice Guidelines, IDH is defined as a decline in systolic blood pressure ≥20 mmHg or a decrease in a mean arterial pressure by 10 mmHg and associated with clinical events like abdominal pain, nausea, vomiting, muscle cramps, dizziness, fatigue, and restlessness.

IDH occurs in response to the reduction in blood volume (BV) during ultrafiltration (UF) and subsequent poor compensatory mechanisms due to abnormal cardiac function (left ventricular dysfunction, chamber remodeling, congenital heart diseases, and arrhythmias) or autonomic or baroreceptor failure. To maintain volume status, the body shifts fluid from the interstitial space to the intravascular space and increases heart rate, contractility, and vascular tone.

Plasma refilling, another essential factor in maintaining euvolemia, depends on oncotic, osmotic, and hydraulic gradients across vascular beds. If UF rates surpass plasma refilling rates, intravascular volume falls and hypotension results. Hematocrit levels, tissue hydration and arterial vasoconstriction all promote plasma refilling rates. Alterations in these factors during dialysis decrease the plasma refilling rate, resulting in hypotension.

Aim of The Work:

The aim of this study is to assess and evaluate the efficacy and safety of L Carnitine in the prevention of intradialytic hypotension in pediatric patients on regular hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 6-18 years
* Patients on hemodialysis for 3 months or longer
* Patients on hemodialysis frequency 3 times weekly (with the same dialysate concentration and temperature)
* Patients who had two or more episodes of intradialytic hypotension during dialysis (less than the 5th percentile of SBP measurements and is associated with clinical symptoms) in the last 3 months.

Exclusion Criteria:

* Patients with life expectancy < 3 months
* Patients with known hypersensitivity to L carnitine
* Patients received L carnitine in the previous 6 months

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-12-10 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
The number of events of intradialytic hypotension | Baseline
  how many times intradialytic hypotension occurs
The number of events of intradialytic hypotension | 3 months (end of the study)
  how many times intradialytic hypotension occurs

SECONDARY OUTCOMES:
development of any adverse effects or side effect in the L carnitine group. | up to 3 months
  monitor the adverse effect that can occur in group 2 due to the drug

CONTACTS AND LOCATIONS:
Locations (1):
- Radwa Maher El Borolossy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No